CLINICAL TRIAL: NCT07061223
Title: Comparative Analysis of the Effectiveness and Safety of Suprainguinal Fascia Iliaca Block (SFIB) and Pericapsular Nerve Group (PENG) Block in the Anesthesia Complex for Total Hip Replacement
Brief Title: SFIB vs PENG Block in the Anesthesia for Total Hip Replacement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSC-02-25
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Regional Anesthesia; Hip Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia with SFIB (Experimental): In this group, under the ultrasound control, a local anesthetic will be injected into the interfacial space of the iliac muscle, in the area of the passage of the deep artery that surrounds the ilium. The block will be performed over the inguinal fold medial to the upper anterior iliac spine. After ultrasound identification of the needle's location in the interfacial space, 40 ml of a 0.5% solution of Ropivacaine will be administered.
  Interventions: Procedure: SFIB; Procedure: Patient control analgesia; Procedure: General inhalation anaesthesia
- General anesthesia with PENG block (Experimental): The block is performed using ultrasound navigation. After identifying the ileo-lumbar tendon, 40 ml of 0.5% Ropivacaine solution is injected under it. Ropivacaine spreads through the hip joint capsule and blocks small sensitive branches of the femoral and obturator nerves.
  Interventions: Procedure: PENG block; Procedure: Patient control analgesia; Procedure: General inhalation anaesthesia
- Control group with general inhalation anesthesia (Other): The control group will undergo general inhalation anesthesia with bolus intraoperative administration of Fentanyl before particularly traumatic stages. For postoperative pain relief, the patient will have the opportunity to use a fentanyl bolus according to the patient-controled analgesia protocol.
  Interventions: Procedure: Patient control analgesia; Procedure: General inhalation anaesthesia

INTERVENTIONS:
Procedure: SFIB — The block technique is based on administration of a local anesthetic under the iliac fascia to block the femoral, lateral femoral cutaneous, and obturator nerves. It is assumed that further leakage of local anesthetic through the interfascial space leads to blocking of the branches of the lumbar plexus in the small pelvis.
  Arms: General anesthesia with SFIB
Procedure: PENG block — The hip capsule is the main source of pain because the innervation of the joint capsule is a developed network of articular branches of the femoral, sciatic and obturator nerves. The main idea of this technique is to block these branches at the point of common passage between the tendon of the lumbar muscle and the crest of the pubic bone. The block technique is based on administration of a local anesthetic under the ileo-lumbar tendon. Anesthetic spreads through the hip joint capsule and blocks small sensitive branches of the femoral and obturator nerves.
  Arms: General anesthesia with PENG block
Procedure: Patient control analgesia — In the postoperative period, if pain occurs, the patient will be offered the opportunity to use 20 ug Fentanyl solution bolus according to the patient control analgesia (PCA) without a basic infusion.
Procedure: General inhalation anaesthesia — General inhalation anesthesia will be performed in all groups, Desflurane with a minimal alveolar concentration (MAC) of 0.6-0.8 will be used for maintenance

SUMMARY:
Total hip replacement is one of the most common orthopedic operations. According to statistical studies, more than 1 million of such surgical interventions are performed annually in the world. The average age of primary hip replacement surgery is 69 y.o.

Modern approaches of control of general anesthesia allow safe performance of different surgical interventions under general anesthesia. However, general anesthesia does not have an effective and long-lasting effect on relieving operational stress compared to neuraxial anesthesia. To achieve a similar effect, it is necessary to adhere to the principle of multimodality of anesthesia, and the most promising method is a combination of general and regional anesthesia. peripheral blocks are described in the literature, aimed at analgesia directly in the hip joint area, and effectively used in orthopedics.

Most blocks are currently performed under ultrasound control, the risk of nerve damage and accidental intravascular administration of local anesthetics is potentially reduced. It was established that the use of ultrasound guidance reduces the number of attempts and the amount of anesthetic administered, as well as reduces the time required to perform a block.

Another predicted effect is a reduction in the doses of opioids and non-steroidal anti-inflammatory drugs (NSAIDs), which can cause gastrointestinal bleeding and have a nephrotoxic effect, and can also depress breathing. It should be noted that patients over 65 y.o., have the highest risks of these side effects.

This study aims to compare the effectiveness and safety of SFIB and PENG block in hip replacement, as well as evaluation of the effectiveness of combined anesthesia in comparison with general anesthesia without the use of peripheral blocks.

DETAILED DESCRIPTION:
Patients will be randomized into three groups group:

Group 1: General anesthesia with SFIB

In this group, under the ultrasound control, a local anesthetic will be injected into the interfacial space of the iliac muscle, in the area of the passage of the deep artery that surrounds the ilium. The block will be performed over the inguinal fold medial to the upper anterior iliac spine. After ultrasound identification of the needle's location in the interfacial space, 40 ml of a 0.5% solution of Ropivacaine will be administered.

Group 2: General anesthesia with PENG block

The block is performed using ultrasound navigation. After identifying the ileo-lumbar tendon, 40 ml of 0.5% Ropivacaine solution is injected under it. Ropivacaine spreads through the hip joint capsule and blocks small sensitive branches of the femoral and obturator nerves.

Group 3: Control group with general inhalation anesthesia

The control group will undergo general inhalation anesthesia with bolus intraoperative administration of Fentanyl before particularly traumatic stages. For postoperative pain relief, the patient will have the opportunity to use a fentanyl bolus according to the patient-controled analgesia protocol.

The following parameters will be evaluated

* Hemodynamic parameters in the intraoperative period
* Intraoperative monitoring of basal metabolic rate using indirect calorimetry
* Monitoring of glucose levels during the most traumatic stages of surgery
* Recording the total dose of opioid analgesics in the perioperative period
* Degree of postoperative pain and analgesic therapy administered
* Block execution time
* Complications of conducting anesthesia
* Degree of patient satisfaction with anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Signed, dated informed consent form
* Age from 50 to 75 years
* Indications for primary total hip replacement
* American Society of Anesthesiologists (ASA) score from 1 to 3

Exclusion Criteria:

* Patients receiving beta blockers;
* Infectious manifestations at the puncture site;
* Bleeding, clinically significant hypovolemia of any origin, shock;
* Disorders of the blood coagulation system;
* Intolerance to local anesthetics;
* Demyelinating diseases of the nervous system;
* Allergy to local anesthetics;
* Psychiatric diseases;
* Any conditions that prevent obtaining informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Total dose of opioid analgesics | 24 hours after surgery
  The total amount of consumed fentanyl required for pain relief will be recorded 24 hours after surgery. For this purpose number of fentanyl boluses will be multiplied on dose size for each included patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 months after completion of the study
Access Criteria: upon the reasonable request